CLINICAL TRIAL: NCT05909982
Title: Effect of Ischemic Post-conditioning on Infarct Volume in Patients With Acute Ischemic Stroke After Mechanical Thrombectomy
Brief Title: Ischemic Post-conditioning in Acute Ischemic Stroke Thrombectomy (PROTECT-1b)
Acronym: PROTECT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTECT-1b
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke; Reperfusion Injury
MeSH Terms: conditions — Ischemic Stroke; Reperfusion Injury | interventions — Ischemic Postconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ischemic post-conditioning group (Experimental): Mechanical thrombectomy combined with ischemic post-conditioning
  Interventions: Procedure: Mechanical thrombectomy combined with ischemic post-conditioning

INTERVENTIONS:
Procedure: Mechanical thrombectomy combined with ischemic post-conditioning — Ischemic post-conditioning will be applied after successful recanalization of the culprit artery by thrombectomy. Ischemic post-conditioning consists of briefly repeated four cycles × 2 minutes of occlusion and reperfusion (equal duration) of the initially occluded artery using a balloon.

SUMMARY:
Ischemic post-conditioning is a neuroprotective strategy attenuating reperfusion injury in animal stroke models. The investigators have conducted a 3 + 3 dose-escalation trial to demonstrate the safety and tolerability of ischemic post-conditioning incrementally for a longer duration of up to 5 min × 4 cycles in stroke patients undergoing mechanical thrombectomy. This study aims to assess the infarct volume after ischemic post-conditioning in patients with acute ischemic stroke who are treated with mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Acute ischemic stroke within 24 hours from stroke onset (or from time last known well) to groin puncture;
* Previous mRS ≤ 2;
* Baseline NIHSS ≥ 6;
* Baseline ASPECTS ≥ 6;
* With an occlusion of unilateral middle cerebral artery M1 segment/distal intracranial carotid artery;
* Successful recanalization (mTICI ≥ 2b) after thrombectomy confirmed by DSA;
* Written informed consent provided by the patients or their legal relatives.

Exclusion Criteria:

* Confirmed or clinically suspected cerebral vasculitis/fibromuscular dysplasia;
* Difficulty in reaching the designated position of the balloon used for ischemic post-conditioning;
* Stenting in the middle cerebral artery M1 segment/distal intracranial carotid artery during thrombectomy;
* > 2 times balloon dilations as rescue therapy due to angioplasty during thrombectomy;
* Moderate/severe residual stenosis (≥ 50%) in the offending artery after thrombectomy;
* Patients with contraindications to MRI;
* Other conditions that the investigator considered inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Infarct volume | 72 hours after procedure
  Infarct volume at 72 hours after procedure

SECONDARY OUTCOMES:
The progression of infarct volume | Baseline and 72 hours after procedure
  Difference of infarct volume between baseline and 72 hours after procedure
The proportion of functional independence at 90 days | 90 days after procedure
  The modified Rankin Scale (mRS) score of 0-2 at 90 days after procedure; the mRS is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
The proportion of favorable outcome at 90 days | 90 days after procedure
  The mRS score of 0-3 at 90 days after procedure; the mRS is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
The distribution of the mRS score at 90 days | 90 days after procedure
  The distribution of the mRS score at 90 days after procedure; the mRS is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
National Institute of Health Stroke Scale (NIHSS) score | 24 hours after procedure
  NIHSS score at 24 hours after procedure; the NIHSS ranges from 0 to 42, with higher scores indicating more severe neurologic deficits
The proportion of early neurological improvement | 24 hours after procedure
  NIHSS 0-2 or ≥8 lower than baseline NIHSS score at 24 hours after procedure; the NIHSS ranges from 0 to 42, with higher scores indicating more severe neurologic deficits
NIHSS score at 7 days after procedure/discharge | 7 days after procedure/discharge
  NIHSS score at 7 days after procedure/discharge; the NIHSS ranges from 0 to 42, with higher scores indicating more severe neurologic deficits
Recanalization rate | 24 hours after procedure
  Recanalization rate at 24 hours after procedure (mTICI ≥2b)
Hemodynamic assessment | Within 24 hours after procedure
  Hemodynamic assessment within 24 hours after procedure

OTHER OUTCOMES:
Safety outcome (mortality at 90 days) | 90 days after procedure
  90-day mortality
Safety outcome (the proportion of symptomatic intracranial hemorrhage within 24 hours) | Within 24 hours after procedure
  The proportion of symptomatic intracranial hemorrhage within 24 hours after procedure
Safety outcome (the proportion of intracranial hemorrhage within 24 hours) | Within 24 hours after procedure
  The proportion of intracranial hemorrhage within 24 hours after procedure
Safety outcome (the proportion of malignant brain edema within 24 hours) | Within 24 hours after procedure
  The proportion of malignant brain edema within 24 hours after procedure
Procedure-related complications | During the procedure
  Vascular perforation/rupture, vessel dissection, severe vasospasm, rupture of the balloon used for post-conditioning

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wu L, Zhang B, Zhao W, Ji X, Wei M. Ischemic post-conditioning in acute ischemic stroke thrombectomy: A phase-I duration escalation study. Front Neurosci. 2022 Dec 8;16:1054823. doi: 10.3389/fnins.2022.1054823. eCollection 2022. PMID 36523440
- [Derived] Jiang X, Wu L, Liu S, Xu Y, Zhang B, Wang S, Luo L, Zhao W, Yao Y, Cao C, Zhao H, Ji X, Wei M. In situ ischemic postconditioning for acute ischemic stroke: preliminary exploratory study. J Neurointerv Surg. 2025 Aug 31:jnis-2025-024031. doi: 10.1136/jnis-2025-024031. Online ahead of print. PMID 40889891